CLINICAL TRIAL: NCT03890289
Title: Idelalisib Plus Obinutuzumab in Patients With Relapsed/Refractory Follicular Lymphoma: a Phase 2, Single-arm, Multicentric Study
Brief Title: Idelalisib+Obinutuzumab in Patients With Relapsed/Refractory Follicular Lymphoma
Acronym: GAUDEALIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted prematurely due to safety, since tocity stopping rules have been met
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_GAUDEALIS
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-07

CONDITIONS: Follicular Lymphoma
Keywords: Idelalisib; Obinutuzumab; Relapsed/Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — idelalisib; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Single arm: Regimen: GAUDEALIS q28 days
  * Obinutuzumab Dose: 1000 mg IV Day 1, 8, 15 (1st cycle)
  * Obinutuzumab Dose: 1000 mg IV Day 1 (2nd cycle onward)
  * Idelalisib Dose: 150 mg BID oral Daily (24 weeks) Obinutuzumab will be administered intravenously at a flat dose of 1000 mg on day 1, 8, 15, of the first cycle, then repeated on day 1 of each subsequent cycle, for 6 cycles in total (each cycle is completed in 28 days). Idelalisib will be given concomitantly with obinutuzumab on a daily 150 mg bid schedule orally and continuously (24 weeks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idelalisib Plus Obinutuzumab (Experimental): Single arm: Regimen: GAUDEALIS q28 days
  * Obinutuzumab Dose: 1000 mg IV Day 1, 8, 15 (1st cycle)
  * Obinutuzumab Dose: 1000 mg IV Day 1 (2nd cycle onward)
  * Idelalisib Dose: 150 mg BID oral Daily (24 weeks)
  Interventions: Drug: Idelalisib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Idelalisib — Idelalisib Plus Obinutuzumab In Patients With Relapsed/Refractory Follicular Lymphoma
Drug: Obinutuzumab — Idelalisib Plus Obinutuzumab In Patients With Relapsed/Refractory Follicular Lymphoma

SUMMARY:
Single arm, prospective, multi-centric, phase II study. Patients with histologically confirmed follicular lymphoma, in need of a systemic approach and failing (i.e. with refractory disease [no response or response lasting less than 6 months at any previous line of treatment] or with a proven disease relapse) at least 2 previous lines of treatment, including any antibody directed against the CD20 antigen-containing chemotherapy, will undergo a combined chemo-free treatment with obinutuzumab and idelalisib.

DETAILED DESCRIPTION:
Single arm, prospective, multi-centric, phase II study. Patients with histologically confirmed follicular lymphoma, in need of a systemic approach and failing (i.e. with refractory disease [no response or response lasting less than 6 months at any previous line of treatment] or with a proven disease relapse) at least 2 previous lines of treatment, including any antibody directed against the CD20 antigen-containing chemotherapy, will undergo a combined chemo-free treatment with obinutuzumab and idelalisib.

Obinutuzumab will be administered intravenously at a flat dose of 1000 mg on day 1, 8, 15 of the first cycle, then repeated on day 1 of each subsequent cycle, for 6 cycles (each cycle is completed in 28 days). Idelalisib will be given concomitantly with obinutuzumab and on a daily 150 mg bid schedule. For patients achieving at least a partial response at the end of induction, a maintenance phase with obinutuzumab is scheduled (on day 1 every two months for two years or until progression or unacceptable toxicity, whichever comes first) If one of the two drugs has to be permanently discontinued due to any cause, patient may continue treatment with the other agent if it is judged to be a clinical benefit. Patients with at least a stable disease will enter the follow-up phase and will be followed with repeated CT scans every six months for two years or until death/progression occurs (whichever comes firsts).

Patients with progressive disease, whenever progression is documented, will enter a survival follow up period of two years after PD was documented. These patients are however considered evaluable for OS.

ELIGIBILITY:
Inclusion criteria

Relapsed or refractory, histologically confirmed CD20-positive follicular non-Hodgkin's lymphoma, grade 1, 2 or 3a according to WHO 2017 classification.

* Age 18 ≥ years
* At least 2 prior systemic therapies for follicular lymphoma including both any antibody directed against the CD20 antigen and a chemotherapy combination.
* Treatment indications, with the presence of at least one of the following:

  * bulky disease (nodal or extranodal mass - except spleen -more than 7 cm in its greater diameter or involvement of at least 3 nodal or extranodal sites, each with a diameter equal to or greater than 3 cm);
  * at least one B-symptom (fever > 38°C of unclear etiology, night sweats, weight loss greater than 10% of body weight in the prior 6 months);
  * symptomatic splenomegaly;
  * compression syndrome (i.e. of orbits, ureters, gastrointestinal tract, biliary tract);
  * lymphoma-related cytopenias (hemoglobin < 10 g/dL and/or platelets < 100.000/mmc and/or neutrophils < 1.500/mmc);
  * pleural or peritoneal serous effusions;
  * lactate dehydrogenase elevation.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
* Adequate hematological function, unless abnormalities due to underlying disease, within 28 days prior to signing informed consent, defined as follows: neutrophils > 1.500/mmc, platelets > 75.000/mmc, hemoglobin > 8,0 g/dL with transfusion independence.
* Capacity and willingness to adhere to study visit schedule and specific protocol procedures.
* Willingness to sign a written informed consent.
* Compliance with effective contraception without interruption, from 28 days before treatment start up (i.e., during the screening phase) to 18 months after treatment discontinuation, agreeing not to donate the semen during treatment and for 18 months after discontinuation (if the patient is male), or to undergo ongoing pregnancy test during the course of the study (if the patient is female).
* Patients must agree to undergo JPJ prophylaxis throughout the treatment period and 2-6 months thereafter (before consulting with Medical Monitor).

Exclusion criteria

Grade 3b follicular non-Hodgkin's lymphoma or evidence of transformation to high-grade non-Hodgkin's lymphoma.

* Central nervous system or leptomeningeal involvement by lymphoma.
* Major surgery (excluding any lymph node biopsy) within 28 days prior to signing informed consent.
* Seropositivity for HBV or evidence of active infection (HBsAg positivity, or HBsAg negativity with positive anti-HBs/anti-HBc and detectable viral DNA load); if viral load is negative or undetectable, the patient is eligible, provided their HBsAg negativity.
* Positive viral HCV RNA
* Seropositivity for HIV, regardless of viral load.
* Known history of drug induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension
* Known history of drug induced pneumonitis
* On-going inflammatory bowel disease
* On-going alcohol or drug addiction
* Life expectancy lower than 6 months.
* Prior history of malignancies, other than follicular lymphoma, unless the patient has been free for at least 10 years (exceptions: localized non-melanoma skin cancer ad carcinoma in situ of the cervix).
* Any of the following laboratory abnormalities: liver enzymes (AST/SGOT and/or ALT/SGPT) > 2.5-fold the upper limit of normal (except of liver involvement by lymphoma); total bilirubin > 1.5 mg/dL (except for patients with known Gilbert's disease or biliary tree compression by lymphoma masses); creatinine clearance < 30 mL/min.
* Uncontrolled intercurrent illness.
* Known hypersensitivity or allergy to murine products or to any of the medicaments under investigation.
* Pregnancy or breastfeeding, or unwillingness to comply with adequate contraception.
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the patient from signing the informed consent or which may place the patient at unacceptable risk if participating in the study.
* Any evidence of ongoing bacterial, viral and fungal infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Zinzani, Prof., Principal Investigator — Bologna - Policlinico S.Orsola-Malpighi - Istituto di Ematologia "Seragnoli"
Locations (4):
- Italy (4):
  - Policlinico S.Orsola-Malpighi - Istituto di Ematologia "Seragnoli", Bologna
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - Azienda sanitaria-universitaria integrata Trieste (ASUITS) - SC Ematologia, Trieste

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Idelalisib Plus Obinutuzumab: Single arm: Regimen: GAUDEALIS q28 days
  * Obinutuzumab Dose: 1000 mg IV Day 1, 8, 15 (1st cycle)
  * Obinutuzumab Dose: 1000 mg IV Day 1 (2nd cycle onward)
  * Idelalisib Dose: 150 mg BID oral Daily (24 weeks)
  Idelalisib: Idelalisib Plus Obinutuzumab In Patients With Relapsed/Refractory Follicular Lymphoma
  Obinutuzumab: Idelalisib Plus Obinutuzumab In Patients With Relapsed/Refractory Follicular Lymphoma
Period: Overall Study
Arm/Group | Idelalisib Plus Obinutuzumab
Started | 5
Completed | 1
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 69 [63 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Ann Arbor Stage [Number; unit: units on a scale] — Ann Arbor staging: better status Stage I, worse status Stage IV.
  units on a scale
    Stage I-II | 0
    Stage III-IV | 5
ECOG Performance Status [Number; unit: units on a scale] — ECOG Performance Status scale: 0 better status, 5 worse status (dead)
  units on a scale
    ECOG 0-1 | 5
    ECOG >1 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint - Overall Response Rate (ORR)
Description: Investigator's assessed Overall response rate at the end of induction phase of patients treated with a chemo-free combination with obinutuzumab and idelalisib. Overall response rate is defined as the proportion of patients with at least a partial response according with 2014 Lugano criteria.
Time Frame: Six months after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Participants
  ORR (CR+PR) | 3
  SD/PD | 2

2. Secondary Outcome: Secondary Endpoints 1 - Overall Survival (OS) Rate
Description: Overall survival (OS) rate, measured from the date of starting therapy to the date of death from any cause. Patients alive and patients who are lost to follow up at the time of the final analysis will be censored at the date of the last contact.
Time Frame: Up to 24 months from the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Participants
  Alive when stopped the study | 4
  Death | 1

3. Secondary Outcome: Secondary Endpoints 2 - Progression-free Survival (PFS) Rate
Description: Progression-free survival (PFS) rate: measured from the date of starting therapy to the date of disease progression, relapse or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last assessment date. Patients who will have no tumor assessment after the start of therapy due to interruption of both drugs will be considered failures at the date of treatment interruption in the PFS analysis
Time Frame: Up to 24 months from the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Participants
  Progression or death any cause when stop the study | 3
  No events when stop the study | 2

4. Secondary Outcome: Secondary Endpoints 3 - Patients' Withdrawal Rate
Description: patients' withdrawal rate, incidence and nature of any severe adverse events hospitalization rate throughout the study, and patients' compliance to oral treatment, incidence of any adverse events occurring during and right after treatment
Time Frame: Up to 24 months from the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Participants
  Early withdrawal along induction | 4
  Not wthdrawed in induction | 1

5. Other Pre Specified Outcome: Safety Monitoring
Description: In order to monitor the safety of the treatment in small cohorts of patients, the Bayesian approach of Thall, et al. for monitoring toxicity will be used. We have planned the monitoring of toxicity to ensure that the proportion of patients with non-hematological toxicity defined as any non-hematological toxicity of grade 3 or higher after 3 and 6 cycles of induction was not higher than an acceptable level of 25%. The prior probability of toxicity (25%) is modeled by a beta distribution [Beta (0.5,1.5)].
Time Frame: Six months from start of treatment
Population: Safety monitoring analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib Plus Obinutuzumab
Number analyzed (Participants) | 5
Participants
  No relevant toxicity | 2
  Relevant toxicity | 3

ADVERSE EVENTS:
Time Frame: Recorded from first dose of study drug through 30 days after the last dose of treatment: about 2.5 years
Arm/Group | Idelalisib Plus Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib Plus Obinutuzumab (N=5)
Pyrexia, respiratory failure, cough (General disorders) | 1 (2)
Pyrexia, diarrhea, Cytomegalovirus reativation (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib Plus Obinutuzumab (N=5)
Fever (General disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (General disorders) | 3 (3)
Transaminasis (Gastrointestinal disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Sars-COV-2 (Infections and infestations) | 1 (1)
CMV reativation (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03890289/Prot_SAP_000.pdf